CLINICAL TRIAL: NCT00101855
Title: Parent Initiated Prevention Program
Brief Title: Can Parental Activation Over the Internet Improve Pediatric Preventive Care?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HS013302-03 (AHRQ)
Record Dates: First submitted 2005-01-14; First posted 2005-01-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-01

CONDITIONS: Well Child Preventive Care
Keywords: prevention; internet; quality of care

INTERVENTIONS:
Procedure: An evidence based tailored web site

SUMMARY:
This study is a randomized controlled trial of an evidence based, patient specific web site's ability to improve preventive practices in pediatric care. Parents visit the website within 2 weeks of a scheduled well child visit and are presented with a menu of age specific topics that they can read about as they wish.

ELIGIBILITY:
Inclusion Criteria:

* <11 years

Exclusion Criteria:

* Non-English speaking

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000
Dates: Start 2003-10; Study Completion 2006-06

PRIMARY OUTCOMES:
Prevention Practices
Satisfaction with care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States